CLINICAL TRIAL: NCT05030493
Title: Additional Exploratory Analysis of Biomarkers in the PARADIGM Exploratory Study in Patients With Advanced/Recurrent Colorectal Cancer
Brief Title: An Additional Analysis of Data From the PARADIGM Exploratory Study (NCT02394834) in Patients With Advanced/Recurrent Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Panitumumab-4006; jRCT1031210293 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P; mFOLFOX6 + panitumumab combination therapy: OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 panitumumab: 6 mg/kg mFOLFOX6 + panitumumab combination therapy, once every two weeks
  Interventions: Drug: mFOLFOX6 + panitumumab combination therapy
- Group B; mFOLFOX6 + bevacizumab combination therapy: OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 bevacizumab: 5 mg/kg mFOLFOX6 + bevacizumab combination therapy, once every two weeks
  Interventions: Drug: mFOLFOX6 + bevacizumab combination therapy

INTERVENTIONS:
Drug: mFOLFOX6 + panitumumab combination therapy — oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab oxaliplatin (OXA), levofolinate calcium (l-LV), panitumumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Groups: Group P; mFOLFOX6 + panitumumab combination therapy
Drug: mFOLFOX6 + bevacizumab combination therapy — oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, bevacizumab oxaliplatin (OXA), levofolinate calcium (l-LV), bevacizumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Groups: Group B; mFOLFOX6 + bevacizumab combination therapy

SUMMARY:
The main aim of the study is to check gene change in tumor tissues with an additional analysis of the data from PARADIGM Exploratory Study, which is conducted for people with advanced/recurrent colorectal cancer.

In the PARADIGM Exploratory Study (NCT02394834), the drug being tested in this study is called Panitumumab and the main aim of this study is to check side effect from the study treatment (mFOLFOX6 + bevacizumab versus mFOLFOX6 + panitumumab therapy) and check if the study treatment improves symptoms of advanced/recurrent colorectal cancer.

DETAILED DESCRIPTION:
This is a non-interventional study to do additional exploratory analysis of biomarkers from the PARADIGM Exploratory Study (NCT02394834), which is conducted for participants with advanced/recurrent colorectal cancer. 757 patients have enrolled in the PARADIGM Exploratory Study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants enrolled in the PARADIGM Exploratory Study (NCT02394834) who have consented to the secondary use of samples and genomic data and have not withdrawn their consent.
2. Participants with sufficient surplus samples for gene expression/mutation and pathomorphologic (IHC, IF and/or ISH, etc.) analysis.

Exclusion Criteria:

Participants who are considered inappropriate for participation in this study by the research institution.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in the PARADIGM Exploratory Study (NCT02394834) who have consented to the secondary use of samples and genomic data and have not withdrawn their consent.
Sampling Method: Probability Sample
Enrollment: 787 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 63 months
  OS obtained in the main study will be stratified by the gene expression levels in tumor tissues at the baseline of the main study to evaluate the relationship between OS and gene expression. OS will be measured as the time from the date of randomization to the date of death due to any causes.
Progression-Free Survival (PFS) | Up to approximately 63 months
  PFS obtained in the main study will be stratified by the gene expression levels in tumor tissues at the baseline of the main study to evaluate the relationship between the PFS and gene expression. PFS is defined as the time from the date of randomization to the earlier of Progressive Disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Evaluation of Correlation between Each Gene Mutations in Plasma Free DNA at Baseline of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months
Evaluation of Correlation between Each Gene Expression Levels in Tumor Tissue at Baseline of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months
Evaluation of Correlation between Change in Each Gene Mutations in Plasma Free DNA at Baseline and Discontinuation of Protocol Treatment of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months
Evaluation of Correlation between Change in Each Gene Expression Levels in Tumor Tissue at Baseline and Discontinuation of Protocol Treatment of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months
Evaluation of Correlation between High Gene Expression Region in Tumor Tissue at Baseline of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months
Evaluation of Correlation between Change in Gene Expression Region in Tumor Tissue at Baseline and Discontinuation of Protocol Treatment of Main Study, and Efficacy Endpoints (OS and PFS) | Up to approximately 63 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/613825d1c61629002b6311e7